CLINICAL TRIAL: NCT04719520
Title: Efficiency Analysis of Wireless Vibrating Caller Compared With Traditional Broadcasting in Contacting Patients' Family Members During Surgery
Brief Title: Efficiency Analysis of Wireless Vibrating Caller During Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202010016RINA
Record Dates: First submitted 2021-01-17; First posted 2021-01-22 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Communication
Keywords: Operating room; Telecommunication experts
MeSH Terms: conditions — Communication

STUDY DESIGN:
Intervention Model Description: This study is a comparative study of the benefits of different ways of contacting patients' family members during surgery.
Masking Description: This study is a comparative study of the benefits of different ways of contacting patients' family members during surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional method (No Intervention): radio and telephone to notify the patient's family to the operating room
- wireless vibrating caller (Experimental): using the wireless vibrating caller to notify the patient's family to the operating room
  Interventions: Behavioral: wireless vibrating caller

INTERVENTIONS:
Behavioral: wireless vibrating caller — using the wireless vibrating caller to notify the patient's family to the operating room
  Arms: wireless vibrating caller

SUMMARY:
As the number of operation increases, it is important to control of the utilization rate of the operating room. This study is a comparative study of the benefits of different ways of contacting patients' family members during surgery.

DETAILED DESCRIPTION:
As the number of operation increases, it is important to control of the utilization rate of the operating room. When family members need to be contacted during the operation, whether family members in the waiting area can be notified in time will affect the overall operation time of the patient and the utilization rate of the operating room. The way of contact also indirectly affects issues such as hospital costs and patient privacy. This study is a comparative study of the benefits of different ways of contacting patients' family members during surgery.

This study will compare the current traditional method (using radio and telephone to notify the patient's family to the operating room) or the wireless vibrating caller to notify the patient's family to the operating room, and analyze the variables generated by the two different methods including demand time of notification, acceptance, and patient privacy issues. The results of the study will use scientific data to prove which way to notify the patient's family is more efficient and a good way to take into account of the patient's privacy.

ELIGIBILITY:
Inclusion criteria:

* The care family of surgical patients

Exclusion criteria:

.The surgical patient's care family has the problems of impaired hearing activity or walking disability.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
demand time | 1 day
  demand time of notifying the patient's family

SECONDARY OUTCOMES:
acceptance | 1 day
  Questionnaire to assess the acceptance the notifying system by the patient's family

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Ming Huang, MD, Ph.D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan